CLINICAL TRIAL: NCT00917332
Title: Effects of Relaxation and Guided Imagery Training on Rate and Time of Receiving Regional Anesthesia (Epidural), and on the Experience of Childbirth
Brief Title: Effects of Relaxation and Guided Imagery Training on Pain at Childbirth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: david mankuta MD, hadassah ein-kerem - obstetrics and gynecology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0256-09-HMO
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Pain at Childbirth
Keywords: pain; childbirth; relaxation; guided imagery; VAS; epidural
MeSH Terms: conditions — Pain | interventions — Respiration; Imagery, Psychotherapy

ARMS (2):
- intervention (Experimental): 55 third trimester women will receive a CD of relaxation and guided imagery (of "safe place"), to practice daily at home until childbirth
  Interventions: Behavioral: relaxation (breathing and muscles) and guided imagery ("safe place")
- control (No Intervention): 55 third trimester women who does not receive the relaxation and guided imagery CD.

INTERVENTIONS:
Behavioral: relaxation (breathing and muscles) and guided imagery ("safe place") — intervention group: daily practice of relaxation and guided imagery CD, for a rew weeks, until childbirth.
  Arms: intervention

SUMMARY:
The purpose of this study is to determine whether relaxation and guided imagery techniques are effective in reducing childbirth pain.

ELIGIBILITY:
Inclusion Criteria:

* women who carry their first child
* women that carry only one embryo
* women who speaks hebrew

Exclusion Criteria:

* women who experienced complications in pregnancy.
* women who planning on having an elective Caesarean section.
* women who suffer from background systematic condition (such as high-BP, diabetes).
* women who have psychiatric background.
* women who take chronic medication that might effect childbirth, woman or baby's health.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-10 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
rating of pain experienced during childbirth on pain VAS | one time - during hospitalization after childbirth

SECONDARY OUTCOMES:
rate and the starting time of receiving regional anesthesia (epidural) | at childbirth

CONTACTS AND LOCATIONS:
Overall Officials: david mankuta, MD, Principal Investigator — hadassah ein-kerem - obstetrics and gynecology
Locations (1):
- Hadassah Ein-Kerem Haspitol, Jerusalem, Israel